CLINICAL TRIAL: NCT04071483
Title: Correlation of Intravascular Injection Rate and Severity of Cervical Neural Foraminal Stenosis During Cervical Transforaminal Epidural Steroid Injection: a Prospective Study
Brief Title: Correlation of Intravascular Injection Rate and Severity of Cervical Neural Foraminal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2018-06-009-001
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Analgesia, Epidural
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate stenosis (Experimental): Moderate cervical neural foraminal stenosis is narrowest width of the neural foramen was >50% of the width of the width of the extraforaminal nerve root at the level of the anterior margin of the superior articular process.
  Interventions: Procedure: Cervical transforaminal epidural steroid injection
- Severe stenosis (Active Comparator): Severe cervical neural foraminal stenosis is narrowest width of the neural foramen was ≤50% of the extraforaminal nerve root width
  Interventions: Procedure: Cervical transforaminal epidural steroid injection

INTERVENTIONS:
Procedure: Cervical transforaminal epidural steroid injection — Cervical transforaminal epidural steroid injection is a useful option in the diagnosis and treatment of cervical radicular pain.

SUMMARY:
This study evaluates whether there is a correlation between intravascular injection rate and severity of cervical foraminal stenosis during cervical transforaminal epidural steroid injection

DETAILED DESCRIPTION:
Cervical transforaminal epidural steroid injection (CTFESI) is useful option to improve cervical radicular pain. However, severe complication can occur by CTFESI such as epidural hematomas, infection, inadvertent intramedullary cord injections, and embolic infarct when inadvertent intra-arterial injection of particulate steroids has occurred.

The incidence of intravascular injection during CTFESI was known as 20.6% ~ 32.8% and it is higher than other level of spinal transforaminal epidural injection.

To avoid complication due to intravascular injection during CTFESI, risk factors was should be evaluated. However, there was no study about risk factors of intravascular injection during CTFESI. The investigators could assume the severity of cervical neural foraminal spinal stenosis could affect the incidence of intravascular injection, pain intensity and effectiveness during CTFESI.

Thus, the investigators designed this study to investigate whether there is a correlation between intravascular injection rate and severity of cervical foraminal stenosis during CTFESI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiating pain from cervical spinal stenosis and herniated nucleus pulposus.

Exclusion Criteria:

* Pregnancy, allergic to contrast media, patient refusal, and patients with persistent contraindication to nerve block such as coagulopathy and infection of the injection site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Intravascular injection | During procedure
  Intravascular injection is defined as contrast media spreading out through the vascular channel during injection of contrast media under real time fluoroscopy

SECONDARY OUTCOMES:
Pain intensity | Before treatment and at 1 month after treatment
  Pain intensity will be evaluated using a numeric rating scale (NRS) from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea